CLINICAL TRIAL: NCT02988466
Title: Reduced Intensity (RIC) Conditioning And Transplantation of HLA-Haploidentical Related Hematopoietic Cells (Haplo-HCT) For Patients With Hematologic Malignancies
Brief Title: Reduced Intensity (RIC) Conditioning And Transplantation of HLA-Haplo-HCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS092; MT2016-15 (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Malignancies
Keywords: Acute Leukemias; Acute myeloid leukemia (AML); Acute lymphoblastic leukemia (ALL)/lymphoma; Biphenotypic/Undifferentiated/Prolymphocytic Leukemias; Myelodysplastic syndrome; Chronic myelogenous leukemia; Minimal Residual Disease (MRD) positive leukemia; Leukemia or Myelodysplastic Syndromes (MDS) in aplasia; Myeloproliferative neoplasms/myelofibrosis; Relapsed large-cell lymphoma, mantle-cell lymphoma and Hodgkin lymphoma; Burkitt's lymphoma; Relapsed T-cell lymphoma; Natural Killer cell malignancies; Relapsed chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, follicular lymphoma; Lymphoplasmacytic lymphoma; Relapsed multiple myeloma; Bone marrow failure syndromes
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasm, Residual; Leukemia; Myeloproliferative Disorders; Primary Myelofibrosis; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, T-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Multiple Myeloma; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Haplo-HCT <55 years old (Experimental): Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients <55 years old with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≤2
  Interventions: Biological: Haplo HCT <55 years old; Drug: GVHD Prophylaxis
- CLOSED Arm B: Haplo-HCT ≥55 years old (Experimental): Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients ≥55 years old or younger with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≥3.
  Interventions: Biological: Haplo HCT ≥55 years old; Drug: GVHD Prophylaxis
- Arm C: Haplo-HCT HCT-CI ≤2 aged ≥55 and < 65yo (Experimental): Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≤2 aged ≥55 and < 65 years old.
  Interventions: Drug: GVHD Prophylaxis; Biological: Haplo HCT ≥55 and < 65 years old
- Arm D: Haplo-HCT aged ≥65 and ≤75yo OR any age HCT-CI ≥3 (Experimental): Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients patients ≥65 and ≤75 years old OR any age group with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≥3.
  Interventions: Drug: GVHD Prophylaxis; Biological: Haplo HCT ≥65 and ≤75 years old

INTERVENTIONS:
Biological: Haplo HCT <55 years old — * Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Melphalan (Mel)
  * Total body irradiation (TBI)
  * Non-T-cell depleted donor bone marrow stem cell infusion Day 0
  Other Names: HLA-haploidentical related hematopoietic cells transplant
  Arms: Arm A: Haplo-HCT <55 years old
Biological: Haplo HCT ≥55 years old — * Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Melphalan (Mel): Dose reduction by 30%
  * Total body irradiation (TBI)
  * Non-T-cell depleted donor bone marrow stem cell infusion
  Other Names: HLA-haploidentical related hematopoietic cells transplant
  Arms: CLOSED Arm B: Haplo-HCT ≥55 years old
Drug: GVHD Prophylaxis — * Cyclophosphamide (Cy)
  * Tacrolimus (Tac)
  * Mycophenolate mofetil (MMF)
Biological: Haplo HCT ≥55 and < 65 years old — * Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Melphalan (Mel)
  * Total body irradiation (TBI)
  * non-T-cell depleted donor bone marrow stem cells
  Other Names: HLA-haploidentical related hematopoietic cells transplant
  Arms: Arm C: Haplo-HCT HCT-CI ≤2 aged ≥55 and < 65yo
Biological: Haplo HCT ≥65 and ≤75 years old — * Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Total body irradiation (TBI)
  Other Names: HLA-haploidentical related hematopoietic cells transplant
  Arms: Arm D: Haplo-HCT aged ≥65 and ≤75yo OR any age HCT-CI ≥3

SUMMARY:
This is a single institution phase II study of a reduced intensity conditioning (RIC) followed by a haploidentical hematopoietic cell transplant (haplo-HCT) in persons with diagnosis of hematologic malignancy. Conditioning will consists of fludarabine, cyclophosphamide, melphalan and total body irradiation (TBI) preparative regimen with a melphalan dose reduction for patients ≥55 years old and those with HCT Comorbidity Index (CI) >3. This study uses a two-stage phase II design with accrual goal of 84 patients, using 28 patients separately for arms A, C and D

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status of ≥70% or Lansky play score ≥ 70%
* A related haploidentical bone marrow donor with up to 2 or 3 HLA locus-mismatches
* The donor and recipient must be HLA identical for at least one haplotype (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1.
* Adequate liver and renal function
* Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction ≥ 40%
* Diffusion capacity corrected (DLCOcorr) > 40% predicted, and absence of O2 requirements
* > 6 months after prior autologous transplant (if applicable)
* Agrees to use contraception during study treatment
* Voluntary written consent (adult or parent/guardian with presentation of the minor information sheet, if appropriate)
* Patients who are HIV+ must have undetectable viral load. All HIV+ patients must be evaluated by Infectious Disease (ID) and a HIV management plan establish prior to transplantation

Exclusion Criteria:

* < 70 years with an available 5-6/6 HLA-A, B, DRB1 matched sibling donor
* Pregnancy or breastfeeding
* Current active and uncontrolled serious infection
* Acute leukemia in morphologic relapse/persistent disease defined as > 5% blasts in normocellular bone marrow OR any % blasts if blasts have unique morphologic markers (e.g. Auer rods).
* CML in blast crisis
* Large cell lymphoma, mantle cell lymphoma and Hodgkin disease that is progressive on salvage therapy.
* stable non-bulky disease is acceptable.
* Active central nervous system malignancy

Criteria For Donor Selection:

* Donors must be HLA-haploidentical relatives of the patient, defined as having a shared HLA haplotype between donor and patient at HLA-A, -B, -C, and -DRB1.
* Eligible donors (14-70 years old) include biological children, siblings or half siblings, or parents, able and willing to undergo bone marrow harvesting.
* For donors <18 years, the maximum recipient weight (actual body weight) should not exceed 1.25 times the donor weight (actual body weight)1 In addition, bone marrow product volume should be limited to 20 ml/kg donor weight for donors <18 years.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2025-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Haplo-HCT <55 Years Old: Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients <55 years old with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≤2
  Haplo HCT <55 years old: - Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Melphalan (Mel)
  * Total body irradiation (TBI)
  * Non-T-cell depleted donor bone marrow stem cell infusion Day 0
  GVHD Prophylaxis: - Cyclophosphamide (Cy)
  * Tacrolimus (Tac)
  * Mycophenolate mofetil (MMF)
- CLOSED Arm B: Haplo-HCT ≥55 Years Old: Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients ≥55 years old or younger with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≥3.
  Haplo HCT ≥55 years old: - Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Melphalan (Mel): Dose reduction by 30%
  * Total body irradiation (TBI)
  * Non-T-cell depleted donor bone marrow stem cell infusion
  GVHD Prophylaxis: - Cyclophosphamide (Cy)
  * Tacrolimus (Tac)
  * Mycophenolate mofetil (MMF)
- Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo: Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≤2 aged ≥55 and < 65 years old.
  GVHD Prophylaxis: - Cyclophosphamide (Cy)
  * Tacrolimus (Tac)
  * Mycophenolate mofetil (MMF)
  Haplo HCT ≥55 and < 65 years old: - Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Melphalan (Mel)
  * Total body irradiation (TBI)
  * non-T-cell depleted donor bone marrow stem cells
- Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3: Reduced-intensity conditioning and transplantation of human leukocyte antigen (HLA) -haploidentical related donor stem cells for patients patients ≥65 and ≤75 years old OR any age group with hematopoietic cell transplantation Comorbidity Index (HCT-CI) ≥3.
  GVHD Prophylaxis: - Cyclophosphamide (Cy)
  * Tacrolimus (Tac)
  * Mycophenolate mofetil (MMF)
  Haplo HCT ≥65 and ≤75 years old: - Fludarabine (Flu)
  * Cyclophosphamide (Cy)
  * Total body irradiation (TBI)
Period: Overall Study
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
Started | 14 | 21 | 8 | 35
Completed | 9 | 10 | 2 | 21
Not Completed | 5 | 11 | 6 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3 | Total
Number analyzed (Participants) | 14 | 21 | 8 | 35 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 8 | 11 | 48
  >=65 years | 0 | 6 | 0 | 24 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 12 | 31
  Male | 8 | 13 | 3 | 23 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 14 | 18 | 8 | 32 | 72
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 1 | 5
  White | 10 | 16 | 5 | 31 | 62
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 14 | 21 | 8 | 35 | 78

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Percentage of participants that were disease-free survival (DFS) at 1 year post-transplant
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
Number analyzed (Participants) | 14 | 21 | 8 | 35
percentage of participants | 57 [28 to 78] | 29 [12 to 48] | 38 [9 to 67] | 57 [39 to 72]

2. Secondary Outcome: Incidence of Grade II-IV and Grade III-IV Acute Graft Versus-host-disease (GVHD)
Description: Percentage of participants with incidence of grade II-IV and grade III-IV acute graft versus-host-disease (GVHD).
Time Frame: day 100
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
Number analyzed (Participants) | 14 | 21 | 8 | 35
Percentage of participants
  grade II-IV acute graft versus-host-disease (GVHD) | 21 [1 to 42] | 33 [13 to 54] | 13 [0 to 34] | 31 [16 to 47]
  grade III-IV acute graft versus-host-disease (GVHD) | 0 [0 to 100] | 19 [3 to 36] | 0 [0 to 100] | 11 [1 to 22]

3. Secondary Outcome: Treatment Related Mortality (TRM)
Description: Percentage of participants experiencing treatment related mortality (TRM).
Time Frame: 6 month, 1 and 2 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
Number analyzed (Participants) | 14 | 21 | 8 | 35
Percentage of participants
  TRM 6 months | 21 [1 to 42] | 57 [39 to 75] | 13 [0 to 34] | 26 [13 to 38]
  TRM 1 year | 21 [1 to 42] | 57 [35 to 79] | 13 [0 to 34] | 26 [11 to 40]
  TRM 2 years | 21 [1 to 42] | 58 [36 to 81] | 13 [0 to 34] | 27 [12 to 42]

4. Secondary Outcome: Relapse Incidence
Description: Percentage of participants experiencing a relapse incidence at 1 and 2 years.
Time Frame: 1 and 2 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
Number analyzed (Participants) | 14 | 21 | 8 | 35
Percentage of participants
  Relapse Incidence 1 year | 29 [5 to 52] | 29 [11 to 46] | 75 [43 to 100] | 26 [11 to 40]
  Relapse Incidence 2 year | 29 [5 to 52] | 30 [11 to 49] | 75 [39 to 100] | 28 [12 to 43]

5. Secondary Outcome: Incidence of Serious Fungal and Viral Infection
Description: Percentage of participants experiencing incidence of serious fungal and viral infection post-HCT
Time Frame: at day 100 and 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
Number analyzed (Participants) | 14 | 21 | 8 | 35
Percentage of participants
  Day 100 | 7 [0 to 20] | 10 [0 to 22] | 38 [6 to 60] | 6 [0 to 13]
  1 year | 14 [0 to 32] | 10 [0 to 22] | 38 [6 to 69] | 11 [1 to 22]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm A: Haplo-HCT <55 Years Old | CLOSED Arm B: Haplo-HCT ≥55 Years Old | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3
All-Cause Mortality (participants affected / at risk) | 6/14 | 13/21 | 5/8 | 18/35
Serious Adverse Events (participants affected / at risk) | 6/14 | 9/21 | 4/8 | 11/35
Other Adverse Events (participants affected / at risk) | 10/14 | 11/21 | 6/8 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Haplo-HCT <55 Years Old (N=14) | CLOSED Arm B: Haplo-HCT ≥55 Years Old (N=21) | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo (N=8) | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3 (N=35)
Serious bacterial Infection (Infections and infestations) | 6 (56) | 9 (133) | 4 (36) | 11 (109)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Haplo-HCT <55 Years Old (N=14) | CLOSED Arm B: Haplo-HCT ≥55 Years Old (N=21) | Arm C: Haplo-HCT HCT-CI ≤2 Aged ≥55 and < 65yo (N=8) | Arm D: Haplo-HCT Aged ≥65 and ≤75yo OR Any Age HCT-CI ≥3 (N=35)
Fungal Infection (Infections and infestations) | 2 (17) | 2 (51) | 3 (22) | 4 (27)
Viral Infection (Infections and infestations) | 9 (95) | 10 (152) | 6 (43) | 12 (67)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT02988466/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT02988466/ICF_001.pdf